CLINICAL TRIAL: NCT00900809
Title: Phase I Study of Adoptive Immunotherapy Using the Natural Killer Cell Line, Neukoplast™(NK-92), for the Treatment of Refractory or Relapsed Acute Myeloid Leukemia
Brief Title: QUILT-3.018: Neukoplast™ (NK-92) for the Treatment of Refractory or Relapsed Acute Myeloid Leukemia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: ImmunityBio, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: QUILT-3.018
Record Dates: First submitted 2009-05-11; First posted 2009-05-13 (Estimated); Last update posted 2022-04-05 (Actual); Status verified 2017-03

CONDITIONS: Acute Myeloid Leukemia
Keywords: Acute Myeloid Leukemia; Neukoplast™; NK-92; Refractory; Refractory or Relapsed Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Neukoplast™ (NK-92) (Experimental): Neukoplast™ will be infused in three doses.1 x 10e9 cells/m2 dose, 3 x 10e9 cells/m2 dose, 5 x 10e9 cells/m2 dose.
  Interventions: Biological: Neukoplast™ (NK-92)

INTERVENTIONS:
Biological: Neukoplast™ (NK-92) — The Neukoplast™ (NK-92) cells will be administered intravenously over 60 minutes. The starting dose of Neukoplast™ (NK-92) cells will be 1 x 10e9 ZRx-101 cells/m2 (The 3 dose levels are: 1 x 10e9 cells/m2, 3 x 10e9 cells/m2 and 5 x 10e9 cells/m2). The second infusion will only be administered after 24 hours if no unacceptable or dose limiting toxicities side effects due to the infusion of Neukoplast™ were encountered after the first infusion.

SUMMARY:
NK cells from patients with malignant diseases are often functionally impaired. Their function cannot be fully restored through ex vivo expansion and cytokine activation. In addition, the in vivo administration of cytokines not only expands NK cells but expands polyclonal T cells with no tumor specificity and no known effects.

The utilization of Neukoplast™, as a form of adoptive immunotherapy, offers several advantages. Neukoplast™ represents a uniform cell population with a well-characterized immunophenotype, confirmed strong anti-tumor activity and are easy to grow and expand in culture, so that they can be made available in large numbers for therapeutic delivery.

ELIGIBILITY:
Inclusion Criteria:

* Patients with refractory/relapse acute myeloid leukemia. Patients must not have received radiotherapy, chemotherapy (with the exception of hydroxyurea which must be discontinued 72 hours prior to therapy) or biological therapy within the preceding 2 weeks of the planned first Neukoplast™ cell infusion and must have recovered from any adverse events due to prior administered agents
* Assessable disease as measured by laboratory and bone marrow examinations
* Age: Eighteen years or older
* Performance status: ECOG ≤ 2 (Appendix A)
* Serum creatinine < 2 X upper limit of normal
* Aspartate aminotransferase (AST) < 5 X upper limit of normal
* Alanine aminotransferase (ALT) < 5 X upper limit of normal
* Total bilirubin < 3X upper limit of normal
* Activated partial thromboplastin time (PTT) < 2.5 X upper limit of normal
* Patients must have left ventricular ejection fraction (LVEF) ≥45 %
* Females of child-bearing potential must have a negative pregnancy test and all subjects must agree to use an effective method of contraception for up to two weeks after the last infusion of Neukoplast™
* Ability to give informed consent
* Life expectancy of greater than 3 months

Note: as many of eligible patients will be pancytopenic secondary to their disease or prior therapies hematologic abnormalities will not be used as a criteria for entry or exclusion.

Exclusion Criteria:

* Patients with acute promyelocytic leukemia
* Symptomatic central nervous system (CNS) involvement
* History of congestive heart failure
* Evidence of severe or uncontrolled systemic diseases (e.g., unstable or uncompensated respiratory, hepatic, renal, or cardiac disease).
* Uncontrolled, life-threatening infection that is not responding to antimicrobial therapy
* ECOG performance status >2 (Appendix A)
* Hepatitis B or C or HIV positive serology
* History of psychiatric disorder which may compromise compliance with the protocol or which does not allow for appropriate informed consent
* Patient may not be receiving any other investigational agents
* Patient is receiving systemic anticoagulation (e.g., warfarin, intravenous heparin. Low dose prophylactic anticoagulation is allowed )
* Patient undergone autologous or allogeneic stem cell transplantation
* Concurrent malignancy of solid tumors. Exception: Subjects who have been disease-free for 5 years, or subjects with a history of completely resected non-melanoma skin cancer or successfully treated in situ carcinoma are eligible. Subjects with second malignancies that are indolent or definitively treated may be enrolled.
* Pregnant or lactating female.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2014-05-12 (Actual); Primary Completion 2015-06-02 (Actual); Study Completion 2015-06-02 (Actual)

PRIMARY OUTCOMES:
Determine the safety / maximum tolerated dose of Neukoplast™ (NK-92 cell line for clinical use) in patients with refractory or relapsed acute myeloid leukemia | 2016

SECONDARY OUTCOMES:
Evaluate the therapeutic efficacy of Neukoplast™ in patients with refractory or relapsed acute myeloid leukemia | 2016
Determine the Neukoplast™ cell phenotype and cytotoxic activity at different time intervals after the Neukoplast™ cell infusion | 2016
Determine the presence of Neukoplast™ in the bone marrow | 2016
Determine the effects of Neukoplast™ on the host immune system, using flow cytometry and the LUMINEX multianalytic profiling system, at different time intervals after the Neukoplast™ infusion. | 2016

CONTACTS AND LOCATIONS:
Overall Officials: Michael Boyiadzis, MD, Principal Investigator — University of Pittsburgh Medical Center
Locations (1):
- UPMC Cancer Center - Hillman Cancer Center, Pittsburgh, Pennsylvania, United States